CLINICAL TRIAL: NCT02743195
Title: An Open Label Study to Investigate a Polyphenol/Prebiotic Blend on Microbial Composition in Otherwise Healthy Obese Males and Females
Brief Title: Polyphenol/Prebiotic Blend Effects on GI Health and Microbial Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 16-PHX-0001; 16PMHN (Other: KGK Synergize Inc.)
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: GI Health; Microbial Composition
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polyphenol/prebiotic blend (Other): Nutritional Supplement. Active ingredients include: Inulin, Fructooligosaccharides, Polyphenol blend of anthocyanin sources--Blueberry extract, Black Currant extract, Black Rice extract. Participants will be instructed to consume one sachet of powder product every morning with breakfast by mixing into beverage or food of choice.
  Interventions: Dietary Supplement: Polyphenol/prebiotic blend

INTERVENTIONS:
Dietary Supplement: Polyphenol/prebiotic blend

SUMMARY:
The gastrointestinal (GI) ecosystem is a complex network of bacterial cells, host cells and tissues that change with age. Fewer numbers and less diversity of beneficial bacteria and greater number and diversity of non-beneficial bacteria occurs with age and conditions associated with accelerated aging (i.e. obesity, high fat diet)(1,2). This imbalance of the microbiota contributes to increased inflammation of the gastrointestinal lining and changes to the integrity of the intestinal cell wall.

Prebiotics, such as non-digestible carbohydrates, can induce the growth or activity microorganisms that contribute to the well-being of the host. Recent studies have shown that prebiotic treatment can have beneficial effects on glucose levels, lipid metabolism, and inflammatory markers in an obese population(3). The polyphenol blend is rich in anthocyanins, which is a unique subgroup of flavonoids that have been demonstrated to impact the microbiome and have anti-inflammatory properties(4,5,6,7). This open-label study will assess the benefits of a prebiotic and polyphenol blend in healthy obese adults.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females 20-60 years of age
2. Female subjects of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

   Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)

   Double-barrier methods

   Non-hormonal intrauterine devices

   Vasectomy of partner

   Non-heterosexual lifestyles
3. Subjects with BMI of 29.9-39.9±1 kg/m²
4. Subjects who agree to maintain their current level of physical activity throughout the trial period
5. Subjects who agree to discontinue the use or pre- and probiotic and/or polyphenol supplements from four weeks prior to baseline and for the duration of the study
6. Subjects who agree to discontinue foods containing anthocyanins (such as blueberries, blackberries, cherries, grapes, grape juice, pomegranate, raspberries, huckleberries, strawberries, and wine) from two weeks prior to baseline and for the duration of the study
7. Healthy as determined by laboratory results and medical history
8. Subjects must agree to comply with study procedures
9. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
2. Subjects who have used an over-the-counter or prescription laxative medication within 4 weeks prior to baseline
3. Subjects who have used prebiotic, probiotic supplements or supplemented foods within 4 weeks of enrollment
4. Use of polyphenol supplements within 4 weeks prior to baseline
5. Subjects with type I diabetes or uncontrolled type II diabetes
6. Previous history of gastrointestinal surgery (except appendectomy, hernia repair, or hemorrhoidectomy).
7. Previous history of gastrointestinal diseases (except hemorrhoids and uncomplicated diverticula), as assessed by ultrasonography, colonoscopy, or rectoscopy, or history of Clostridium difficile-associated diarrhea
8. Presence of rectal bleeding (unless due to hemorrhoids)
9. Recent weight-loss (greater than 5 kg in the past month)
10. Iron deficiency (anemia) diagnosed within 3 months of baseline
11. Subjects who were smokers within 1 year of baseline
12. Subjects with active eating disorder
13. Subjects who have used oral antibiotics within 5 weeks of baseline
14. Unstable medical condition as determined by principal investigator
15. History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years of diagnosis are acceptable.
16. Alcohol abuse or drug abuse within the past 6 months
17. Consumption of >2 standard alcoholic drinks per day
18. Use of medicinal marijuana
19. Use of anti-inflammatory medications, more than once per week or if prescribed by a physician, 4 weeks prior to randomization and for the duration of the study
20. Participation in a clinical research trial within 30 days prior to baseline
21. Allergy or sensitivity to the test material's active or inactive ingredients
22. Allergy or sensitivity to Lactulose or Mannitol
23. Individuals who are cognitively impaired and/or who are unable to give informed consent
24. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in microbial composition in the feces at day 57 | Baseline, Day 57

SECONDARY OUTCOMES:
Change from baseline in calprotectin in the feces at day 57 | Baseline, Day 57
Change from baseline in IL-6 in the feces at day 57 | Baseline, Day 57
Change from baseline in IL-8 in the feces at day 57 | Baseline, Day 57
Change from baseline in IL-10 in the feces at day 57 | Baseline, Day 57
Change from baseline in IL-1β in the feces at day 57 | Baseline, Day 57
Change from baseline in IL-12p70 in the feces at day 57 | Baseline, Day 57
Change from baseline in TNFα in the feces at day 57 | Baseline, Day 57
Change from baseline in urine sugar test for gut permeability at day 57 | Baseline, Day 57
Change from baseline in plasma zonulin at day 57 | Baseline, Day 57
Change from baseline in Total Cholesterol at day 57 | Baseline, Day 57
Change from baseline in HDL-C at day 57 | Baseline, Day 57
Change from baseline in LDL-C at day 57 | Baseline, Day 57
Change from baseline in Triglycerides at day 57 | Baseline, Day 57
Change from baseline in weekly mean of daily Bristol Stool Scale (BSS) scores at day 57 | Baseline, Day 57
Change from baseline in plasma endotoxin at day 57 | Baseline, Day 57

OTHER OUTCOMES:
Change from baseline in hematology and clinical chemistry at day 57 | Baseline, Day 57
  Looking at number of participants with abnormal laboratory values related to treatment
Change from baseline in kidney and liver function at day 57 | Baseline, Day 57
  Looking at number of participants with abnormal laboratory values related to treatment
Change from baseline in electrolytes at day 57 | Baseline, Day 57
Change from baseline in heart rate at day 57 | Baseline, Day 57
Change from baseline in blood pressure at day 57 | Baseline, Day 57
Change from baseline in adverse events at day 57 | Baseline, Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biagi E, Nylund L, Candela M, Ostan R, Bucci L, Pini E, Nikkila J, Monti D, Satokari R, Franceschi C, Brigidi P, De Vos W. Through ageing, and beyond: gut microbiota and inflammatory status in seniors and centenarians. PLoS One. 2010 May 17;5(5):e10667. doi: 10.1371/journal.pone.0010667. PMID 20498852
- [Background] Duncan SH, Flint HJ. Probiotics and prebiotics and health in ageing populations. Maturitas. 2013 May;75(1):44-50. doi: 10.1016/j.maturitas.2013.02.004. Epub 2013 Mar 11. PMID 23489554
- [Background] Everard A, Cani PD. Diabetes, obesity and gut microbiota. Best Pract Res Clin Gastroenterol. 2013 Feb;27(1):73-83. doi: 10.1016/j.bpg.2013.03.007. PMID 23768554
- [Background] Karlsen A, Retterstol L, Laake P, Paur I, Bohn SK, Sandvik L, Blomhoff R. Anthocyanins inhibit nuclear factor-kappaB activation in monocytes and reduce plasma concentrations of pro-inflammatory mediators in healthy adults. J Nutr. 2007 Aug;137(8):1951-4. doi: 10.1093/jn/137.8.1951. PMID 17634269
- [Background] Vendrame S, Guglielmetti S, Riso P, Arioli S, Klimis-Zacas D, Porrini M. Six-week consumption of a wild blueberry powder drink increases bifidobacteria in the human gut. J Agric Food Chem. 2011 Dec 28;59(24):12815-20. doi: 10.1021/jf2028686. Epub 2011 Nov 18. PMID 22060186
- [Background] Guglielmetti S, Fracassetti D, Taverniti V, Del Bo' C, Vendrame S, Klimis-Zacas D, Arioli S, Riso P, Porrini M. Differential modulation of human intestinal bifidobacterium populations after consumption of a wild blueberry (Vaccinium angustifolium) drink. J Agric Food Chem. 2013 Aug 28;61(34):8134-40. doi: 10.1021/jf402495k. Epub 2013 Aug 19. PMID 23883473
- [Background] Taverniti V, Fracassetti D, Del Bo' C, Lanti C, Minuzzo M, Klimis-Zacas D, Riso P, Guglielmetti S. Immunomodulatory effect of a wild blueberry anthocyanin-rich extract in human Caco-2 intestinal cells. J Agric Food Chem. 2014 Aug 20;62(33):8346-51. doi: 10.1021/jf502180j. Epub 2014 Aug 8. PMID 25075866